CLINICAL TRIAL: NCT03333473
Title: Postpregnancy Family Planning Choices in Public and Private Sectors in Kenya and Indonesia
Acronym: PPFP Choices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Merck for Mothers (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00007462
Record Dates: First submitted 2017-10-25; First posted 2017-11-07 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Post-pregnancy Family Planning; Capacity Building of Healthcare Providers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention will be applied to health facilities in one district in Indonesia and one county in Kenya. The intervention package will work within existing public and private health facilities to strengthen and assess the effectiveness of facility and provider level PPFP service provision and counseling, and expand method choice for women during antenatal, early labor, and post-pregnancy pre-discharge periods. Training within the intervention package include provider-lever PPFP counseling and service provision (PPFP Clinical and Counseling Skills), as well as provider and facility-level leadership management and governance training (Facility-Level Leadership Management and Governance Training).
  Interventions: Behavioral: PPFP Clinical and Counseling Skills; Behavioral: Facility-Level Leadership Management and Governance Training
- Control (No Intervention): The health facilities control district in Indonesia and county in Kenya will continue with their standard counseling and service provision throughout the study period. At the conclusion of the study period, the facilities in these areas will receive the same intervention that Intervention facilities received prior to study startup.

INTERVENTIONS:
Behavioral: PPFP Clinical and Counseling Skills — Facilities will receive whole-site orientations on PPFP basics and skills Through training of trainers, followed by classroom and model-based and clinical-based practice, providers will receive training in PPDP counseling and service provision.
  Arms: Intervention
Behavioral: Facility-Level Leadership Management and Governance Training — The intervention will strengthen leadership management and governance practices required to help managers establish PPFP services at the facility level.
  Arms: Intervention

SUMMARY:
The primary goal of PPFP Choices is to generate actionable evidence that can be used to increase programmatic activities to address post-pregnancy family planning in the public and private-for-profit sectors. The ultimate intent of this investment is to advance and scale up post-pregnancy FP. Programmatic learning will be crucial to understanding what it will take to accelerate post-pregnancy FP in these two countries, and these can later be adapted by other countries with similar settings. Our vision of PPFP Choices can be achieved through the following objectives:

* Objective 1: Establish a comprehensive program implementation framework for the private sector to embrace post-pregnancy FP
* Objective 2: Improve the quality of post-pregnancy FP counseling and service provision in both public and private sectors
* Objective 3: Build evidence and contribute to the literature and programmatic guidance around post-pregnancy FP uptake and continuation in both public and private sectors
* Objective 4: Ensure effective documentation and strategic dissemination which will benefit post-pregnancy FP introduction and scale-up more broadly

DETAILED DESCRIPTION:
PPFP Choices is an operations research study seeking to examine the barriers and facilitators in offering a full range of FP methods in the immediate post-pregnancy period in both the public and private sectors.

Jhpiego will implement the study in two counties in Kenya; Meru and Kilifi, and two districts in Indonesia; Brebes and Batang.

This study will employ a quasi-experimental design with an intervention and control group. Prior to study start-up, the the intervention group will receive a Jhpiego-designed package of interventions designed to advance post-pregnancy FP in both the public and private sectors. These interventions draw on WHO's Programming Strategies for Postpartum Family Planning, as well as Jhpiego's experience and assessments. After the study is completed, the control groups will receive the same intervention. For the study, a mixed method approach will be used; both quantitative and qualitative data will be collected through Client Quantitative Interviews, Client In-Depth interviews, Focus Group Discussions, Key Informant Interviews, and Facility Assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Kenyan postpartum participant (Enrollment starts at ANC):

   1. At least 28 weeks pregnant
   2. Plans to deliver at the study facility
   3. Aged 15-49 years at enrollment
   4. Provides voluntary informed consent
   5. Not planning to relocate in the next 12 months
2. Indonesian postpartum participant (Enrollment starts at L&D):

   1. In the immediate postpartum period (within 72 hours, prior to leaving the health facility),
   2. Reported having attended ANC within her 3rd trimester (28-weeks pregnant and later),
   3. Aged 15-49 years at time of enrollment (Indonesian adolescents aged 15-16 must be married for purposes of the study consent)
   4. Provides voluntary informed consent
   5. Not planning to relocate in the next 12 months
3. Kenyan and Indonesian postabortion participants:

   1. A female in the immediate post-pregnancy treatment phase (within 72 hours in Indonesia, within 48 hours in Kenya, prior to leaving the health facility for treatment of incomplete abortion)
   2. Aged 15-49 years at time of enrollment (Indonesian adolescents aged 15-16 must be married for purposes of the study consent)
   3. Provides voluntary informed consent
   4. Not planning to relocate in the next 6 months

Exclusion Criteria:

1. Refusal to sign consent form for inclusion in the study
2. Post-delivery baby or mother being treated for trauma or in an intensive care unit

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants must be women in the ANC period with a gestational age of 28 weeks or greater [Kenya], in the immediate postpartum period (within 72 hours after childbirth)[Indonesia], or immediately following receipt of postabortion care (within 48 hours [Kenya] or 72 hours [Indonesia]).
Enrollment: 9282 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Quality of PPFP counseling | 3 years
  80% of ANC attendees and women receiving postabortion care receive appropriate PPFP counseling prior to discharge compared to baseline in the comparison group.
Clinical competency of service providers in providing all modern FP methods | 3 years
  100% of service providers in intervention arm of study are deemed competent and retain competencies to provide all modern FP methods to women during postpartum and postabortion periods.

SECONDARY OUTCOMES:
Postpartum uptake of LARCs | 3 years
  50% increase in Long-Acting and Permanent Method use by study participants whose infants are six months old in study intervention sites in Indonesia and 70% increase in LARC use by study participants whose infants are six months old in study intervention sites in Kenya. A change in use of LARCs and other permanent methods of FP by study participants whose infants are six months old, from 10% to 15% in Indonesia and from 6% to 10% in Kenya at intervention facilities over the course of the study
Health facility-level leadership management and governance skills | 3 years
  80% of health facilities in the intervention group show improvement in leadership management and government measured through use of quality improvement approaches
Assessment of individual intervention quality | 3 years
  Using a quality improvement framework, assess individual pieces of the intervention package using multi-level modeling

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Charurat, MBA, MHS, Principal Investigator — Jhpiego
Locations (8):
- Indonesia (8):
  - RSUD Batang, Batang, Central Java
  - RSU QOlbu Insan Mulia, Batang, Central Java
  - Puskesmas Subah, Batang, Central Java
  - Puskesmas Bawang, Batang, Central Java
  - RSUD Brebes, Brebes, Central Java
  - Puskesmas Kecipir, Brebes, Central Java
  - Puskesmas Ketanggungan, Brebes, Central Java
  - RSU Alam Medika Bumi Ayu, Brebes, Central Java

IPD SHARING:
Plan to Share IPD: Undecided
The study protocol will be shared through publication in a peer-reviewed journal.
  De-identified participant data will be submitted to a data repository in accordance with the Bill and Melinda Gates Foundation and Merck for Mothers policies.

REFERENCES:
- [Derived] Charurat E, Kennedy S, Qomariyah S, Schuster A, Christofield M, Breithaupt L, Kariuki E, Muthamia M, Kabue M, Omanga E, Stekelenburg J. Study protocol for Post Pregnancy Family Planning Choices, an operations research study examining the effectiveness of interventions in the public and private sectors in Indonesia and Kenya. Gates Open Res. 2020 Dec 18;4:89. doi: 10.12688/gatesopenres.13147.2. eCollection 2020. PMID 33693315

DOCUMENTS (3):
  • Study Protocol (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT03333473/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT03333473/SAP_001.pdf
  • Informed Consent Form (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT03333473/ICF_002.pdf